CLINICAL TRIAL: NCT05833828
Title: Differences in Plasma Concentration of RAAS-axis Hormones in Patients Undergoing Cardiac Surgery With or Without Cardiopulmonary Bypass
Brief Title: Differential Regulation of RAAS-axis in Patients Undergoing Cardiac Surgery
Acronym: RAAS-HLM
Status: Recruiting | Type: Observational
Sponsor: Universität Münster (Other)
Responsible Party: Sponsor
Other Study IDs: AnIt22-08
Record Dates: First submitted 2023-01-19; First posted 2023-04-27 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Vasoplegia; Vasoplegic Shock
Keywords: vasoplegia; vasoplegic shock; cardiopulmonary bypass; cardiac surgery
MeSH Terms: conditions — Vasoplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- on-pump coronary artery bypass graft surgery: Due to the observational design of the study, no study-specific interventions are performed. Except for the above mentioned laboratory analyses, the treatment of the patients is completely guided by the responsible ICU physicians.
  Study participation does not influence the determination of surgical procedure (on- vs off-pump).
  Interventions: Procedure: on-pump surgery
- off-pump coronary artery bypass graft surgery: Due to the observational design of the study, no study-specific interventions are performed. Except for the above mentioned laboratory analyses, the treatment of the patients is completely guided by the responsible ICU physicians.
  Study participation does not influence the determination of surgical procedure (on- vs off-pump).
  Interventions: Procedure: off-pump surgery

INTERVENTIONS:
Procedure: on-pump surgery — the surgery will be performed "on-pump"
  Groups: on-pump coronary artery bypass graft surgery
Procedure: off-pump surgery — the surgery will be performed "off-pump"
  Groups: off-pump coronary artery bypass graft surgery

SUMMARY:
This study investigates the question of whether there are differences in the plasma concentration of hormones of the RAAS-axis between patients undergoing on-pump cardiac surgery and those receiving off-pump surgery

DETAILED DESCRIPTION:
In patients undergoing cardiac surgery, the occurrence of vasoplegia or vasoplegic shock is a common and sometimes very severe complication. Although there are multiple factors that may affect the incidence and severity of vasoplegia, it remains unclear which role the use of cardiopulmonary bypass may play in the pathogenesis of this complication. The heart normally pumps blood through the lungs where the blood primarily gets oxygenated. However, it is also known that pulmonary blood flow is also essential for the activation of various hormones, some of which are central to the regulation of vascular tension and blood pressure. If the pulmonary circulation is bypassed, as is the case in on-pump cardiac surgery, it is likely that the resulting differential activity of hormones may cause or contribute to the incidence of vasoplegia. This study aims to show whether cardiopulmonary bypass leads to the differential regulation of hormones of the renin-angiotensin-aldosterone-system which could explain why some patients suffer from vasoplegia or vasoplegic shock following such procedures.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients undergoing on- or off-pump coronary artery bypass graft surgery
2. written informed consent

Exclusion Criteria:

1. emergency surgery in the context of acute coronary syndrome
2. ACE-inhibitor or Angiotensin 1 (AT1)-receptor-blocker intake that was not paused on the day of surgery
3. Chronic kidney disease with estimated glomerular filtration rate (eGFR)<30ml/min/1.73m²
4. Severe structural lung disease (asbestosis, silicosis, severe sarcoidosis, tuberculosis, severe emphysema, chronic obstructive pulmonary disease (COPD) Gold 3-4, lung fibrosis)
5. Chronic pulmonary hypertension
6. Pregnancy or breastfeeding
7. Persons with any kind of dependency on the investigator or employed by the institution responsible or investigator
8. Persons held in an institution by legal or official order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Differences in plasma concentration of Angiotensinogen | between induction of anesthesia and immediately after surgical intervention
Differences in plasma concentration of Renin | between induction of anesthesia and immediately after surgical intervention
Differences in plasma concentration of Angiotensin I | between induction of anesthesia and immediately after surgical intervention
Differences in plasma concentration of Angiotensin converting enzyme (ACE) | between induction of anesthesia and immediately after surgical intervention
Differences in plasma concentration of Angiotensin II | between induction of anesthesia and immediately after surgical intervention
Differences in plasma concentration of Aldosterone | between induction of anesthesia and immediately after surgical intervention

SECONDARY OUTCOMES:
Differences in plasma concentration of Angiotensin 1-9 | between induction of anesthesia and immediately after surgical intervention
Differences in plasma concentration of Angiotensin 2-7 | between induction of anesthesia and immediately after surgical intervention
Differences in plasma concentration of Dipeptidyl-peptidase 3 (DPP3) | between induction of anesthesia and immediately after surgical intervention
Incidence of vasoplegia | within 12 hours post surgery
Cumulative dose of vasopressors | within 12 hours post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zarbock, MD, Study Chair — University Hospital Muenster, Dept. of Anesthesiology, Intensive Care Therapy and Pain Medicine
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum der Charité, Berlin
  - University Hospital Münster; Department of Anesthesiology, Intensive Care Medicine and Pain Medicine, Münster

IPD SHARING:
Plan to Share IPD: No